CLINICAL TRIAL: NCT05761977
Title: Durvalumab in Combination With Standard Chemotherapy for 1st Line Therapy of Patients With Extensive Stage Small Cell Lung Cancer: A Non-interventional, Prospective Observational Study of Clinical Practice, Quality of Life and Use of Health Resources in Real-world Clinical Practice (DRIVE)
Brief Title: Durvalumab in Combination With Standard Chemotherapy of Patients With Extensive Stage Small Cell Lung Cancer
Acronym: DRIVE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: HE1R/21
Record Dates: First submitted 2023-02-07; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Small-cell Lung Cancer; Extensive-stage Small-cell Lung Cancer
Keywords: observational study; small- cell lung cancer; extensive-stage small-cell lung cancer; first line treatment
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with extensive small-cell lung cancer: extensive small-cell lung cancer

SUMMARY:
This is a non-interventional, multicenter, prospective observational study and registry of standard clinical practice in patients with Extensive Stage-Small Cell Lung Cancer (ES-SCLC) receiving 1st line treatment with Durvalumab in combination with standard chemotherapy (cisplatin or carboplatin + etoposide) in the approved indication, which will be carried out in Greece. In this study data will be collected prospectively based on real-world clinical practice. A prospective cohort of atients from centers of the Hellenic Cooperative Oncology Group (HeCOG) will be included. The study will be conducted in hospitals and by physicians specialized in lung cancer from different geographical areas of Greece.

DETAILED DESCRIPTION:
In this observational prospective study, no changes to current therapeutic practice will be required and all aspects of treatment and clinical management of patients will be in compliance with the local clinical practice and will be left to the discretion of the participating physicians. Patients will be treated in accordance with the study medicine's local prescribing information and standard clinical practice as to the frequency of visits and types of evaluations carried out. The frequency of follow-up visits is set on the basis of standard practice; however, the study-related data will be collected during integration and during the routine clinical visits that will take place after the start of treatment. No visits or measurement/evaluation will be mandatory by the protocol and data collection at the predetermined time-points will be carried out only if the patient visits the center.

Patients will be enrolled during a 12-month recruitment period from HeCOG-participating public and private centers/clinics in Greece with specialization in lung cancer. As part of this study, participating physicians will be asked to follow up each patient for an additional 12 months of treatment at most after last subject is included, or until death, withdrawal of consent, discontinuation of treatment or initiation of new antineoplastic therapy, until completion of the study, or doctor's decision, whichever appears first. Therefore, the maximum period of prospective observation of the study will be 24 months (2 years) from the last patient enrolled in the study. This study will be conducted in accordance with the Guidelines for Good Pharmacoepidemiological Practice, the European General Data Protection Regulation (GDPR) and the applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, regardless of race (residents in Greece), no younger than 18 years old at the initiation of treatment.
* Patients with histologically or cytologically confirmed diagnosis of extensive Small Cell Lung Cancer (SCLC)
* Patients who have not received prior systemic treatment for SCLC (chemotherapy or immunotherapy)
* Patients for whom the decision to administer treatment with Durvalumab+chemotherapy has already been taken before their inclusion in the study and is clearly separated from the decision of the physician for the patient's participation in the current study.
* Patients who have provided informed signed consent to participate in the study and to collect and analyze medical data related to the objectives of this study.

Exclusion Criteria:

* Patients with current diagnosis of primary cancer other than SCLC who require systemic or other treatment.
* Patients who have previously received chemotherapy or immunotherapy for SCLC
* Patients who are currently receiving or are expected to receive treatment with an investigational drug/medical device/intervention or who have received an investigational medicinal product within 1 month or 5 years half-life of the research agent (whichever is longer) before their initiation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Small- Cell Lung Cancer candidates for 1st- line immunotherapy plus platinum based chemotherapy (cisplatin or carboplatin plus etoposide) currently with active disease.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival rates (OS) | up to 24 months
  The primary objective of the study is to estimate the overall survival rates (OS) at 6,12 and 24 months for patients with extensive small-cell lung cancer treated with Durvalumab in combination with standard 1st-line chemotherapy with platinum-etoposide(cisplatin or carboplatin).

SECONDARY OUTCOMES:
Progression free survival (PFS) | in 6, 12 and up to 24 months
  Evaluation of PFS from investigator
Overall response rate (ORR) | in 6 and up to 12 months
Disease Control Rate | in 6 and up to 12 months
time to reach a response (TTR) | up to 12 months
duration of the response (DoR) | up to 12 months
Assessment of patients characteristics with overall survival 12 months | up to 12 months
Assessment of patients characteristics with overall survival 24 months | up to 24 months
time under treatment (ToT) | up tp 24 months
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 with standard of care 1st line treatment | From date of Informed Consent signatory and every 3 weeks, up to 24 months
Quality of life EQ-5D | From date of Informed Consent signatory and every 2 months, up to 24 months
number of participants using health resources in daily clinical practice | From date of Informed Consent signatory and every 3 weeks, up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Helena Linardou, MD, Principal Investigator — Metropolitan Hospital of Athens
Locations (1):
- Metropolitan Hospital, Neo Faliro, Greece

IPD SHARING:
Plan to Share IPD: No